CLINICAL TRIAL: NCT05613088
Title: A Phase 2 Open-label Randomized Study of Farletuzumab Ecteribulin (MORAb-202), a Folate Receptor Alpha-targeting Antibody-drug Conjugate, Versus Investigator's Choice Chemotherapy in Women With Platinum-resistant High-grade Serous (HGS) Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study of MORAb-202 Versus Investigator's Choice Chemotherapy in Female Participants With Platinum-resistant High-grade Serous (HGS) Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA116-001; 2021-004807-42 (EudraCT Number)
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms, Ovarian
Keywords: Platinum-resistant ovarian cancer (PROC); Primary peritoneal cancer; Fallopian tube cancer; MORAb-202; Folate-receptor alpha; ADC; Antibody-drug conjugate; Epithelial ovarian cancer; High grade serous; Farletuzumab ecteribulin
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — MORAb-202; Paclitaxel; liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MORAb-202 (Experimental)
  Interventions: Drug: MORAb-202
- Investigator's Choice Chemotherapy (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Topotecan

INTERVENTIONS:
Drug: MORAb-202 — Specified dose on specified days
  Other Names: BMS-986445; Farletuzumab Ecteribulin
  Arms: MORAb-202
Drug: Paclitaxel — Specified dose on specified days
  Other Names: Bendalis
  Arms: Investigator's Choice Chemotherapy
Drug: Pegylated Liposomal Doxorubicin (PLD) — Specified dose on specified days
  Other Names: Caelyx
  Arms: Investigator's Choice Chemotherapy
Drug: Topotecan — Specified dose on specified days
  Other Names: Hycamtin
  Arms: Investigator's Choice Chemotherapy

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and efficacy of farletuzumab ecteribulin (MORAb-202) and compare it to Investigator's choice (IC) chemotherapy in female participants with platinum-resistant HGS ovarian, primary peritoneal, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with histologically-confirmed diagnosis of HGS ovarian, primary peritoneal, or fallopian tube cancer.
* Platinum-resistant disease, defined as:
* For participants who had only 1 line of platinum-based therapy: progression between > 1 month and ≤ 6 months after the last dose of platinum-based therapy of at least 4 cycles.
* For participants who had 2 or 3 lines of platinum-based therapy: progression ≤ 6 months after the last dose of platinum-based therapy.
* Participants have received at least 1 but no more than 3 prior lines of systemic therapy and for whom single-agent therapy is appropriate as the next line of therapy. Participants may have been treated with up to 1 line of therapy subsequent to determination of platinum-resistance.
* Disease progression per RECIST v1.1 (by investigator assessment) of at least 1 measurable lesion on or after the most recent therapy.
* Either formalin-fixed, paraffin-embedded (FFPE) tissue (up to 5 years old) or newly-obtained biopsies must be available for FRα assessment prior to randomization.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.

Exclusion Criteria:

Medical Conditions

* Clear cell, mucinous, endometrioid or sarcomatous histology, or mixed tumors containing components of any of these histologies, or low grade or borderline ovarian cancer.
* Primary platinum-refractory ovarian cancer defined as disease progression within 1 month of the last dose of the first line platinum-containing regimen.
* Pulmonary function test (PFT) abnormalities: FEV1 < 70% or FVC < 60%, and DLCO < 80%.
* Investigator-assessed current ILD/pneumonitis, or ILD/pneumonitis suspected at screening or history of ILD/pneumonitis of any severity including ILD/pneumonitis from prior anti-cancer therapy.
* Significant third-space fluid retention (eg, ascites or pleural effusion) that requires repeated drainage.

Physical and Laboratory Test Findings

* Evidence of organ dysfunction or any clinically-significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population.

Allergies and Adverse Drug Reactions

* Has any prior severe hypersensitivity (≥ Grade 3) to monoclonal antibodies or eribulin or contraindication to the receipt of corticosteroids or any of the excipients (investigators should refer to the prescribing information for the selected corticosteroid).
* History of allergy or contraindication to IC chemotherapy agent selected if randomized to Arm C.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2025-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (50):
- United States (10):
  - Local Institution - 0065, Sacramento, California
  - Local Institution - 0025, San Francisco, California
  - Local Institution - 0078, Whittier, California
  - Local Institution - 0081, South Bend, Indiana
  - Local Institution - 0043, Kansas City, Kansas
  - Local Institution - 0023, Canton, Ohio
  - Local Institution - 0061, Columbus, Ohio
  - Local Institution - 0044, Nashville, Tennessee
  - Local Institution - 0082, Salt Lake City, Utah
  - Local Institution - 0042, Spokane, Washington
- Australia (6):
  - Local Institution - 0016, Sydney, New South Wales
  - Local Institution - 0017, Waratah, New South Wales
  - Local Institution - 0031, Chermside, Queensland
  - Local Institution - 0015, Clayton, Victoria
  - Local Institution - 0027, Malvern, Victoria
  - Local Institution - 0058, Nedlands, Western Australia
- Belgium (4):
  - Local Institution - 0032, Leuven, VBR
  - Local Institution - 0013, Namur, WNA
  - Local Institution - 0012, Brussels
  - Local Institution - 0045, Liège
- Chile (3):
  - Local Institution - 0030, Santiago, RM
  - Local Institution - 0036, Santiago
  - Local Institution - 0029, Temuco
- Israel (5):
  - Local Institution - 0046, Jerusaelm, JM
  - Local Institution - 0054, Haifa
  - Local Institution - 0080, Jerusalem
  - Local Institution - 0055, Ramat Gan
  - Local Institution - 0048, Tel Aviv
- Italy (5):
  - Local Institution - 0003, Bologna, BO
  - Local Institution - 0011, Milan, MI
  - Local Institution - 0009, Milan, MI
  - Local Institution - 0010, Roma, RM
  - Local Institution - 0002, Brescia
- Japan (5):
  - Local Institution - 0018, Akashi, Hyogo
  - Local Institution - 0019, Chūōku
  - Local Institution - 0014, Hidaka-shi
  - Local Institution - 0004, Kurume-Shi
  - Local Institution - 0037, Tokyo
- South Korea (3):
  - Local Institution - 0056, Seoul
  - Local Institution - 0049, Seoul
  - Local Institution - 0053, Seoul
- Spain (9):
  - Local Institution - 0039, Barcelona, B
  - Local Institution - 0005, Madrid, M
  - Local Institution - 0001, Madrid, M
  - Local Institution - 0007, Valencia, V
  - Local Institution - 0006, Valencia, V
  - Local Institution - 0021, Barcelona
  - Local Institution - 0020, Girona
  - Local Institution - 0038, Madrid
  - Local Institution - 0022, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was stopped and no participants were enrolled into Arm A (MORAb-202 at 33 mg/m^2)
Groups:
- MORAb-202: Participants received MORAb-202 25 mg/m^2 every 3 weeks for up to 2 years
- Investigator's Choice (IC) Chemotherapy: Participants received Paclitaxel 80 mg/m^2 every week; OR
  Pegylated liposomal doxorubicin (PLD) 40 mg/m^2 every 4 weeks; OR
  Topotecan 4 mg/m^2 Days 1, 8,15 every 4 weeks or 1.25 mg/m^2 Days 1 to 5 every 3 weeks for up to 2 years
Period: Pre-Treatment
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Started (Started = Randomized) | 70 | 36
Completed (Completed = Treated) | 70 | 34
Not Completed | 0 | 2
Period: Treatment
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Started (Started = Treated) | 70 | 34
Completed | 0 | 0
Not Completed | 70 | 34
Not completed — Ongoing Study Treatment | 9 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Other Reasons | 0 | 1
Not completed — Progressive Disease | 58 | 26
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy | Total
Number analyzed (Participants) | 70 | 36 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (9.15) | 61.3 (12.16) | 59.3 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 36 | 106
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 57 | 29 | 86
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 50 | 24 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Per Investigator Assessment
Description: Objective Response Rate (ORR) is defined as the number of randomized participants who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on investigator assessments [using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1], divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to the date of first objectively-documented progression or the date of subsequent therapy (Up to approximately 70 weeks)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 36
Percent of participants | 20.0 [11.4 to 31.3] | 13.9 [4.7 to 29.5]

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Event (TRAEs) Leading to Discontinuation Within 6 Months From First Dose
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after starting study treatment, whether or not considered related to the study intervention.
Time Frame: From first dose of study medication up to 6 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 2 | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: as for outcome 2
Time Frame: From the first dose of study medication until 17Jun2024, which is 30 days after the last dose of study treatment (assessed for an average duration of approximately 5 months, with a maximum of up to 14 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 67 | 32

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 19 | 10

5. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation
Description: as for outcome 2
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 3 | 0

6. Secondary Outcome: Number of Participants With Treatment-Related AEs
Description: as for outcome 2
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 53 | 29

7. Secondary Outcome: Number of Participants With Treatment-Related SAEs
Description: as for outcome 4
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 1 | 2

8. Secondary Outcome: Number of Participants With AEs of Special Interest (AESIs)
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after starting study treatment, whether or not considered related to the study intervention.
  AEs of special interest include: Infusion-related reactions, Interstitial lung disease (ILD) and Pneumonitis
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants
  Infusion-related reactions | 1 | 1
  Interstitial lung disease (ILD) | 2 | 0
  Pneumonitis | 13 | 0

9. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died during the study.
Time Frame: From first dose of study medication until death due to any cause (up to 70 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants | 21 | 6

10. Secondary Outcome: Number of Participants With Grade 3-4 Laboratory Abnormalities
Description: Number of participants experiencing clinical abnormalities in laboratory testing including hematology, chemistry, liver function, and renal function.
  Laboratory findings are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 34
Participants
  Grade 3: Lymphocytes (absolute) | 3 | 0
  Grade 3: Absolute neutrophil count | 3 | 9

11. Secondary Outcome: Disease Control Rate (DCR) by RECIST v1.1 Per Investigator Assessment
Description: Disease Control Rate (DCR) is defined as the number of randomized participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD), based on investigator assessments (using RECIST v1.1) divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  Based on Clopper and Pearson estimates of duration of response
Time Frame: From the date of randomization to the first date of documented progression, or death whichever occurs first (Up to approximately 70 weeks)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 36
Percent of participants | 80.0 [68.7 to 88.6] | 69.4 [51.9 to 83.7]

12. Secondary Outcome: Duration of Response (DoR) by RECIST v1.1 Per Investigator Assessment
Description: Duration of Response (DoR) is defined as the time between the date of first documented response (CR or PR) confirmed, to the date of the first objectively documented tumor progression by investigator (per RECIST v1.1) or death, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates of duration of response
Time Frame: From the date of first dose to the date of the first documented tumor progression, or death, whichever occurs first (Up to approximately 70 weeks)
Population: All confirmed responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 14 | 5
Months | 4.42 [2.50 to NA] — Insufficient number of events for upper limit | 5.55 [2.37 to NA] — Insufficient number of events for upper limit

13. Secondary Outcome: Progression-free Survival (PFS) by RECIST v1.1 Per Investigator Assessment
Description: Progression-free Survival (PFS) is defined as the time between the date of randomization and the first date of documented progression, per investigator assessments (using RECIST v1.1), or death due to any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates of progression-free survival
Time Frame: as for outcome 11
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 70 | 36
Months | 4.01 [2.79 to 4.67] | 4.40 [3.98 to 6.67]
Statistical Analysis 1: Comparison: MORAb-202 vs Investigator's Choice (IC) Chemotherapy; Test type: Superiority; p = 0.4063, Log Rank; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.76 to 2.00]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from randomization until death or data cut off date 29Apr2025 (up to approximately 70 weeks). SAEs and Other AEs from first dose of study medication until 29Apr2025 (up to approximately 70 weeks).
Description: All-cause Mortality refers to all randomized participants. SAEs and other AEs refers to all the participants who were treated with study medicine.
Arm/Group | MORAb-202 | Investigator's Choice (IC) Chemotherapy
All-Cause Mortality (participants affected / at risk) | 34/70 | 18/36
Serious Adverse Events (participants affected / at risk) | 22/70 | 11/34
Other Adverse Events (participants affected / at risk) | 61/70 | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-202 (N=70) | Investigator's Choice (IC) Chemotherapy (N=34)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 5 | 3
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-202 (N=70) | Investigator's Choice (IC) Chemotherapy (N=34)
Anaemia (Blood and lymphatic system disorders) | 10 | 8
Leukopenia (Blood and lymphatic system disorders) | 6 | 3
Neutropenia (Blood and lymphatic system disorders) | 7 | 10
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 15 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 17 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 17 | 15
Stomatitis (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 9 | 5
Asthenia (General disorders) | 12 | 6
Fatigue (General disorders) | 11 | 7
Mucosal inflammation (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 5 | 2
Pyrexia (General disorders) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 3
Alanine aminotransferase increased (Investigations) | 6 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood albumin decreased (Investigations) | 2 | 2
Blood magnesium decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 2 | 9
Platelet count decreased (Investigations) | 0 | 3
Weight decreased (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 14 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 2 | 3
Lymphoedema (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT05613088/Prot_SAP_000.pdf